CLINICAL TRIAL: NCT06607055
Title: Monitoring of Immunity Markers in Intensive Care Patients and Link with Recurrence and Relapse of Ventilator-associated Pneumonia
Brief Title: Immunity Markers in Intensive Care Patients and Ventilator-associated Pneumonia
Acronym: IMMUNAIX
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Aix-Pertuis (Other)
Responsible Party: Principal Investigator, Laurent LEFEBVRE, Principal investigator, Centre Hospitalier Intercommunal Aix-Pertuis
Other Study IDs: 20232704-9
Record Dates: First submitted 2024-08-28; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Pneumonia, Ventilator-Associated
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — HLA-DR dosage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Interventional - blood collection: HLA-DR dosage, at the time of inclusion and once a week then
  Interventions: Diagnostic Test: Blood collection

INTERVENTIONS:
Diagnostic Test: Blood collection — HLA-DR dosage, at the time of inclusion and once a week then

SUMMARY:
The goal of this observational study is to show the direct correlation between the occurrence of recurrence of VAP and postagressive immunoparalysis, monitored by HLA-DR rate below litterature-acknowledged threshold, in a well conducted antibiotherapy context, in patient admitted in the Intensive Care Unit.

The main questions it aims to answer are:

* evaluation of the association between death and persistence of immunoplegia using HLA-DR monitoring
* search an association between immunoplegia depth and severity of the initial state of shock
* search an association between immunoplegia depth and viral reactivation
* compare association of immunoplegia duration and HLA-DR nadir and VAP occurrence Blood samples will be taken from participants to HLA-DR dosage, at the time of inclusion and once a week then.

DETAILED DESCRIPTION:
The occurrence of ICU-acquired infections in patients admitted to the intensive care unit (ICU) results in increased morbidity and mortality, increased length of stay in the ICU, and also clearly increased healthcare costs. The incidence of these infections fluctuates between 15% and 40%, depending on the study. A major problem in the ICU is the recurrence and relapse of ventilator-associated pneumonia (VAP), with increased exposure to antibiotics and a probable increase in average length of stay.

One of the possible hypothesis that could explain relapses/recurrences of VAP is incorrect conducted antibiotherapy. To prevent this, in the unit, we currently perform antibiotics pharmacological assays and adapt them to the antibiogram. Another possible explanation to treatment failure could be patients' postagressive immunoparalysis. It has clearly been demonstrated that postagressive immunoparalysis is a predisposing state to healthcare related infections.

Some markers can be used to monitor this immunoplegia state. Several studies have shown that low HLA-DR expression and reduced CD16 expression (polymorphonuclear neutrophils percentage) is associated with increased susceptibility to develop infections in the ICU.

Immunity monitoring could be an interesting tool to identify populations most at risk of developing healthcare-associated infections after a state of shock, and could become an interesting line of thinking for the use of immunomodulatory therapies. To best evaluate these therapies and find a place for them in the current arsenal, it is essential to integrate them into daily practice by linking them to a significant clinical event, such as recurrent healthcare-associated infections, despite properly conducted antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient admitted in the Intensive Care Unit of the CHIAP
* Patient under mechanical ventilation
* Patient with infectious pneumonia
* Informed Consent Form (ICF) obtained from the patient or emergency ICF obtained from close relatives
* Patient beneficiary of French social security, whatever the regime

Exclusion Criteria:

* Patient under 18 years old
* Patient with severe neutropenia (neutrophils < 0.5 G/L)
* Patient under immunosuppressive treatment
* Use of corticosteroids (intravenous or oral) prior to ICU admission
* Use of therapeutic antibodies
* Onco-hematological disease (e.g. lymphoma, leukemia...) under treatment or treated in the 5 years prior to inclusion
* End of chemotherapy 6 months prior to inclusion
* Patients with innate or acquired immune deficiency (e.g., severe combined immunodeficiency, HIV or AIDS, at any stage)
* Patients with a decision to limit or discontinue active therapies, at the time of inclusion
* Patients with an estimated ICU stay of less than 48 hours
* Participation in an interventional study
* Patient deprived of their liberty
* Patient under tutorship or curatorship
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted in the ICU of the CHIAP under mechanical ventilation and with infectious pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a VAP recurrence/relapse | From date of hospital admission until the date of the end of hospitalization or date of death from any cause, whichever came first, assessed up to 100 months
  Number of occurrence of a VAP recurrence/relapse

SECONDARY OUTCOMES:
Viral reactivation | From date of hospital admission until the date of the end of hospitalization or date of death from any cause, whichever came first, assessed up to 100 months
  To search for association between immunoplegia depth and viral reactivation (CMV)
Association between immunoparalysis depth and state of shock severity within the first 24 hours | First 24 hours
  To search for association between immunoplegia depth and severity of the initial state of shock (lactatemia, amine dosage, SOFA score over 48 hours)
Persistence of immunoparalysis during hospitalization and care-related infections | From date of hospital admission until the date of the end of hospitalization or date of death from any cause, whichever came first, assessed up to 100 months
  To compare association of immunoplegia duration and HLA-DR nadir and VAP occurrence
HLA-DR nadir and link with care-related infections | From date of hospital admission until the date of the end of hospitalization or date of death from any cause, whichever came first, assessed up to 100 months
  To compare association of immunoplegia duration and HLA-DR nadir and VAP occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Laurent LEFEBVRE, MD, Principal Investigator — Centre Hospitalier Intercommunal Aix-Pertuis
Locations (1):
- Centre Hospitalier Intercommunal Aix-Pertuis, Aix-en-Provence, France

IPD SHARING:
Plan to Share IPD: No